CLINICAL TRIAL: NCT04176107
Title: The Effect of Exposure to Informative Video Before Cesarean Delivery on Maternal Anxiety and Peripartum Satisfaction- a Randomized Control Trial
Brief Title: The Effect of Exposure to Informative Video Before Cesarean Delivery on Maternal Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0092-19-WOMC
Record Dates: First submitted 2019-10-22; First posted 2019-11-25 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2019-11

CONDITIONS: Maternal Distress (During Labor); Anxiety
Keywords: Cesarean delivery; Anxiety; Informative-video
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group- video+questionnaire (Other): The study group will be exposed to a video at admission to an elective cesarean delivery. The video will have information regarding the admission, pre-operation preparation and post- operation recovery.
  All patients will answer a questionnaire at admission, before surgery and 24 hours later. the questionnaires will evaluate the impact of exposure to informative video before caesarean delivery on anxiety and stress measured by State-Trait Anxiety Inventory (STAI).
  Interventions: Behavioral: Informative video
- Control group- questionnaire only (No Intervention): All patients will answer a questionnaire at admission, before surgery and 24 hours later. the questionnaires will evaluate anxiety and stress measured by State-Trait Anxiety Inventory (STAI) without intervention.

INTERVENTIONS:
Behavioral: Informative video — Exposure to informative video before cesarean delivery
  Arms: Study group- video+questionnaire

SUMMARY:
The incidence of cesarean deliveries (CD) worldwide is increasing, around 30% in United States. Although very common surgery women undergoing non emergent CD still experience fear and anxiety. It is known that increased levels of stress can negatively affect pain perception and the usage of analgesics postoperatively as well as lactation.

this present study investigate the effect of exposure to informative video before cesarean delivery on maternal anxiety.

DETAILED DESCRIPTION:
A multi-center randomized control trial the will examine the effect of exposure to informative video before cesarean delivery on maternal anxiety and satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Hebrew speaking
* Informed consent
* First cesarean delivery
* Non emergent elective CD

Exclusion Criteria:

* Non Hebrew speaking
* Refuse to participate
* Emergency CD

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 126 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
The State-Trait Anxiety Inventory STAI:Y-1 | Baseline (Questionnaire filled by the patient Before operation)
  Psychological questionnaire to assess stress and anxiety-The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 20 questions on a self-report basis. Higher scores are positively correlated with higher levels of anxiety.

SECONDARY OUTCOMES:
The State-Trait Anxiety Inventory STAI:Y-1 | Questionnaire filled by the patient at admission- 1 day before operation
  Psychological questionnaire to assess stress and anxietyhe State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 20 questions on a self-report basis. Higher scores are positively correlated with higher levels of anxiety.
Childbirth experience questionnaire (CEQ) | Questionnaire filled by the patient at 1 day after the delivery
  Questionnaire to evaluate the women experience and satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: hadas miremberg, MD, Principal Investigator — Wolfson Medical Center
Locations (4):
- Israel (4):
  - Haemek Medical Center, Afula
  - Asuta Medical Center, Ashdod
  - Rambam Medical Center, Haifa
  - Wolfson medical center, Holon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miremberg H, Yirmiya K, Vinter D, Lauterbach R, Yefet E, Nassra R, Paz YG, Hagege R, Weiner E. An informative video before planned cesarean delivery and maternal anxiety-a multicenter randomized controlled trial. Am J Obstet Gynecol MFM. 2022 May;4(3):100604. doi: 10.1016/j.ajogmf.2022.100604. Epub 2022 Feb 28. PMID 35240345